CLINICAL TRIAL: NCT02343224
Title: A Phase II Study Of Pegylated Interferon ALFA-2b in Children With Recurrent or Refractory and Radiographically or Clinically Progressive Juvenile Pilocytic Astrocytomas and Optic Pathway Gliomas
Brief Title: Pegylated Interferon ALFA-2b in Children With Juvenile Pilocytic Astrocytomas and Optic Pathway Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: CURE Childhood Cancer, Inc. (Other)
Responsible Party: Principal Investigator, Dolly Aguilera, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00074563
Record Dates: First submitted 2015-01-08; First posted 2015-01-21 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Juvenile Pilocytic Astrocytomas; Optic Pathway Gliomas
MeSH Terms: conditions — Astrocytoma | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegylated interferon alpha-2b (Experimental): Subjects will receive PEG-Intron based on their weight (1 mcg/kg/dose) once a week
  Interventions: Drug: Pegylated interferon alpha-2b

INTERVENTIONS:
Drug: Pegylated interferon alpha-2b — PEG-Intron 1mcg/kg/dose weekly through an injection under the skin on the same day each week
  Other Names: Peg-Intron

SUMMARY:
This is a phase II study of the drug, pegylated interferon alfa-2b (PEG-Intron), used to treat brain tumors in a pediatric population. Researchers want to see if treatment with PEG-Intron will stop tumor growth for patients with juvenile pilocytic astrocytomas or optic pathway gliomas.

The purposes of this study are:

* To learn more about the response to pegylated interferon
* To learn more about the side effects of pegylated interferon
* To learn more about MRI images in patients with Juvenile Pilocytic Astrocytomas or Optic Pathway Gliomas.
* To learn more about quality of life in patients treated with pegylated interferon

DETAILED DESCRIPTION:
Low grade gliomas are the most common pediatric central nervous system malignancies and can occur in different parts of the brain. Patients who undergo gross total resection, usually those with hemispheric tumors, have an excellent prognosis with surgical resection alone. Patients for whom gross total resection is not achievable have a significant risk of disease progression. Therefore, these patients benefit from adjuvant therapy. Multiple chemotherapy regimens have shown some efficacy in residual tumor, but more than 50% of patients experience recurrences. Radiation has been shown to be an effective therapy in the treatment of these tumors. Because of concerns regarding radiation toxicity especially in young children, and progression despite chemotherapy, novel approaches are needed. This protocol represents an attempt to measure the efficacy and safety of use of pegylated interferon for patients with recurrent, refractory Juvenile Pilocytic Astrocytomas (JPA) or optic pathway gliomas. It provides a different approach to the commonly used treatment modalities. The objectives of this study are to determine the response of children with chemotherapy-refractory progressive JPA or optic pathway gliomas (OPG) to weekly pegylated interferon alpha-2b. The secondary objectives include to better identify the toxicities of weekly pegylated interferon alpha-2b (PEG-Intron™) in pediatric patients with unresectable, refractory, recurrent JPAs or optic pathway gliomas, to evaluate various magnetic resonance imaging techniques for noninvasive monitoring of metabolic and biologic changes in the tumors and to evaluate the quality of life for patients with recurrent, refractory JPAs who receive therapy with pegylated interferon alpha-2b (PEG-Intron™).

The primary end point is to determine the response rate. A two-stage design has been selected to evaluate the response rate. If the treatment demonstrates at least a 25% response rate, the researchers would consider it a promising regimen for further study. A response rate less than 5% is considered evidence of unpromising regimen. Seventeen evaluable pediatric patients with JPA or OPG will be accrued. If at least 3 responders are seen among the 17 patients, this will be considered evidence of a promising response rate for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be older than 3 years and less than or equal to 25 years of age at the time of enrollment
* Patients with neurofibromatosis are eligible
* Histologic confirmation is not required for this if the patient has neurofibromatosis type 1 (NF-1) with MRI findings consistent with optic pathway glioma or JPA. Any other tumors will need histological confirmation, either at the time of diagnosis or at the time of recurrence. The histological diagnosis includes World Health Organization (WHO) grade I JPA
* Patients must have measurable residual disease, defined as tumor that is measurable in two or three perpendicular diameters on MRI. For a lesion to be considered measurable, it must be at least twice the slice thickness on MRI (i.e visible on more than one slice)
* All patients must have a brain MRI with and without contrast (gadolinium) within 30 days prior to study enrollment. All patients with history of spinal or leptomeningeal disease and those patients with symptoms suspicious of spinal disease, must have a spine MRI with contrast (gadolinium) performed within 30 days prior to study enrollment. Lumbar puncture is necessary if there is evidence of tumor dissemination on the MRI of spine
* Performance Level: Karnofsky > or equal to 50% for patients > 10 years of age or Lansky > or equal to 50 for patients < 10 years of age
* Patients must have recovered (to Common Toxicity Criteria (CTC) v.5.0 ≤ Grade 1 unless indicated below) from the acute toxic effects of all prior chemotherapy, immunotherapy prior to entering this study, with the exception of alopecia, weight changes and Grade I or II lymphopenia

  * Must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
  * At least 7 days must have elapsed since the completion of therapy with other biologic agents. For other biologic agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * At least 3 half-lives of the antibody after the last dose of a monoclonal antibody. Specifically for bevacizumab 36 days after the last dose
  * At least 3 weeks from the last surgical resection, prior to start study drug
  * At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * Patients must have had their last fraction of cranial or craniospinal Radiation ≥ 24 months prior to study entry
  * Patients who have received polyinosinic-polycytidylic acid-polylysine-carboxymethylcellulose (Poly-ICLC) are eligible for this trial if all acute Poly-ICLC -related toxicity has resolved
  * Patients must not have received Pegylated interferon previously
* Must not have received growth factor within 2 weeks of entry into this study
* Patients who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior enrollment in the study
* Adequate organ, hematological, renal, and pulmonary function
* If history of depression or psychiatric illness, has to be well controlled with antidepressants and/or under psychiatrist/psychologist care

Exclusion Criteria:

* Patients who are receiving concurrent chemotherapy, or who are currently receiving other investigational chemotherapeutic agents or concurrently receiving radiation
* Patients with a known hypersensitivity to interferon-alpha
* Prior use of Pegylated interferon or interferon
* Less than 2 years since completion of radiation therapy
* Pregnant or breast-feeding females are excluded
* Patients with clinically significant unrelated systemic illness
* Dental braces or prosthesis that interferes with magnetic resonance (MR) imaging
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Patients with a positive history of Hepatitis B or Hepatitis C
* Male patient whose sexual partner(s) are women of childbearing potential who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Patient with diagnosis of Diffuse Intrinsic Pontine Glioma

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolly Aguilera, MD, Principal Investigator — Children's Healthcare of Atlanta/Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Children's Healthcare of Atlanta, in Atlanta, Georgia. Enrollment began November 2014 and all follow up was complete by November 11, 2020.
Groups:
- PEGINTRON: Participants with juvenile pilocytic astrocytomas or optic pathway gliomas receiving PEGINTRON based on their weight (1 mcg/kg/dose) once a week, for up to two years
Period: Overall Study
Arm/Group | PEGINTRON
Started | 9
Completed | 0
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | PEGINTRON
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 11 [5 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Children Responding to Treatment
Description: The objective response of study participants was categorized as complete response, partial response, or stable disease. Determination of tumor response or progression is based on the pre-study baseline scan performed closest to time of study entry. The overall response assessment takes into account response in both target and non-target lesion, and the appearance of new lesions. Complete response is defined as the disappearance of all target lesions and non-target lesions, and no new lesions. Partial response is defined as ≥ 65% decrease in the sum of the products of the three perpendicular diameters of all target lesions, and no development of new lesions. Stable disease is defined as neither sufficient decrease in the sum of the products of the three perpendicular diameters of all target lesions to qualify for partial response, nor sufficient increase in a single target lesion to qualify for progressive disease, as well as no new lesions.
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | PEGINTRON
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 5

2. Secondary Outcome: Number of Participants Meeting Event Free Survival Criteria
Description: Event free survival is the time to treatment failure from the time of study enrollment to tumor progression, tumor recurrence, death from any cause or occurrence of a second malignant neoplasm.
Time Frame: Month 12, Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | PEGINTRON
Number analyzed (Participants) | 9
Participants
  Month 12 | 7
  Month 24 | 7
Statistical Analysis 1: Comparison: PEGINTRON; This Kaplan-Meier estimate is the conditional probability of event-free survival among study participants at 12 and 24 months; Test type: Other; Kaplan-Meier estimate = 76.2, 95% CI 2-sided [52.1 to 100]

3. Secondary Outcome: Number of Participants Meeting Overall Survival Criteria
Description: Overall survival is measured as the time from study enrollment to death from any cause.
Time Frame: Month 12, Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | PEGINTRON
Number analyzed (Participants) | 9
Participants
  Month 12 | 7
  Month 24 | 7
Statistical Analysis 1: Comparison: PEGINTRON; This Kaplan-Meier estimate is the conditional probability of overall survival among participants at 12 and 24 months; Test type: Other; Kaplan-Meier estimate = 75, 95% CI 2-sided [50.3 to 100]

ADVERSE EVENTS:
Time Frame: Data collection for adverse events began at the Baseline (Day 0) study visit and continued through the time when the participant was removed from the study intervention (up to 2 years).
Description: Information on serious adverse events and adverse events that were related to the study treatment were collected.
Arm/Group | PEGINTRON
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEGINTRON (N=9)
Anorexia, grade 3 (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEGINTRON (N=9)
Abdominal pain, grade 1 (Gastrointestinal disorders) | 1
Increased alanine transaminase (ALT), grade 1 (Hepatobiliary disorders) | 5
Decreased absolute neutrophil count (ANC), grade 1 (Blood and lymphatic system disorders) | 1
Anorexia, grade 2 (General disorders) | 1
Increased aspartate aminotransferase (AST), grade 1 (Hepatobiliary disorders) | 2
Constipation, grade 2 (Gastrointestinal disorders) | 1
Cough, grade 1 (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness, grade 1 (General disorders) | 1
Dry skin, grade 1 (Skin and subcutaneous tissue disorders) | 1
Anemia, grade 1 (Blood and lymphatic system disorders) | 4
Dyspepsia, grade 2 (Gastrointestinal disorders) | 1
Fatigue, grade 1 (General disorders) | 1
Headache, grade 1 (General disorders) | 3
Hypermagnesemia, grade 1 (Blood and lymphatic system disorders) | 2
Hypertriglyceridemia, grade 2 (Blood and lymphatic system disorders) | 1
Hyperuricemia, grade 1 (Blood and lymphatic system disorders) | 3
Hypoalbuminemia, grade 1 (Blood and lymphatic system disorders) | 4
Hypocalcemia, grade 1 (Blood and lymphatic system disorders) | 6
Hypokalemia, grade 1 (Blood and lymphatic system disorders) | 3
Hypophosphatemia, grade 1 (Blood and lymphatic system disorders) | 3
Infection, grade 2 (Infections and infestations) | 1
Decreased lymphocyte count, grade 1 (Blood and lymphatic system disorders) | 2
Nausea, grade 1 (General disorders) | 1
Decreased neutrophil count, grade 1 (Blood and lymphatic system disorders) | 3
Pain at injection site, grade 1 (Injury, poisoning and procedural complications) | 1
Decreased platelet count, grade 1 (Blood and lymphatic system disorders) | 3
Right forearm eczema, grade 1 (Skin and subcutaneous tissue disorders) | 1
Vomiting, grade 2 (Gastrointestinal disorders) | 1
Weight loss, grade 2 (General disorders) | 1
Decreased white blood cell count, grade 1 (Blood and lymphatic system disorders) | 6
Increased ALT, grade 2 (Hepatobiliary disorders) | 1
Anemia, grade 2 (Blood and lymphatic system disorders) | 1
Fatigue, grade 2 (General disorders) | 1
Hypophosphatemia, grade 2 (Blood and lymphatic system disorders) | 1
Decreased lymphocyte count, grade 2 (Blood and lymphatic system disorders) | 4
Decreased neutrophil count, grade 2 (Blood and lymphatic system disorders) | 1
Decreased neutrophil count, grade 3 (Blood and lymphatic system disorders) | 2
Decreased platelet count, grade 3 (Blood and lymphatic system disorders) | 1
Decreased white blood cell count, grade 2 (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT02343224/Prot_SAP_000.pdf